CLINICAL TRIAL: NCT01459289
Title: The Psychosocial Effect of Testing Positive for HPV on Hong Kong Chinese Women With Normal Cervical Cytology
Brief Title: Psychosocial Effect of HPV Positivity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Collaborators: Queen Mary Hospital, Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: UW11-327
Record Dates: First submitted 2011-09-15; First posted 2011-10-25 (Estimated); Last update posted 2011-10-25 (Estimated); Status verified 2011-10

CONDITIONS: Human Papillomavirus
MeSH Terms: interventions — Counseling

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- leaflet (Active Comparator)
  Interventions: Other: leaflet
- counseling (Active Comparator)
  Interventions: Other: counseling and leaflet

INTERVENTIONS:
Other: leaflet
  Arms: leaflet
Other: counseling and leaflet
  Arms: counseling

SUMMARY:
The use of HPV testing in cervical screening has raised concerns about the effect of a positive HPV result on women's psychological well being. This is a nested psychosocial study of the COCY trial (IRB No. UW 09-377; PI: Prof Hextan Ngan), with the aim to evaluate the psychosocial impact of HPV positivity on Hong Kong Chinese women and the modulating effects of educational intervention on such impact. Potential participants are identified among those who have joint the COCY trial. Participants will be randomized into two groups, namely the control group or intervention group. The control group participants will receive their smear results and an HPV leaflet by post. The intervention group will receive the leaflet and a counseling session on HPV. Self-administered questionnaires will be used to assess participants' psychological condition at the receipt of the smear results and at two months afterward. It is hypothesized that the level of emotional distress measured at smear result notification will be greater than that at two months afterward for all participants. Furthermore, participants in the intervention group will have lower psychological distress than those in the control group at two months after the receipt of their smear results.

ELIGIBILITY:
Inclusion Criteria:

1. Ethnic Chinese women who have enrolled in the COCY trial, and whose smear results are normal cytology with HPV positivity
2. Women who are willing to attend colposcopy
3. Literate in the Chinese language
4. Have given a verbal consent to participate in this study

Exclusion Criteria:

* Women who are unable to provide a consent to participation.

Ages: 30 Years to 60 Years | Sex: Female
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2011-10; Primary Completion 2013-10 (Estimated); Study Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in anxiety to 6 months | Level of anxiety will be measured at the receipt of cervical smear results, and at 2-months and 6-months afterward.
  Anxiety meausred by the Hospital Anxiety and Depression Scale

SECONDARY OUTCOMES:
Change from baseline in depression to 6 months | Level of depression will be measured at the receipt of cervical smear results, and at 2-months and 6-months afterward.
  Depression will be measured by the Hospital Anxiety and Depression Scale

CONTACTS AND LOCATIONS:
Overall Officials: Hextan YS Ngan, MD, Principal Investigator — The University of Hong Kong
Locations (1):
- Department of Obstetrics & Gynaecology, The University of Hong Kong, Hong Kong, China